CLINICAL TRIAL: NCT05585541
Title: Comparison of the International Cooperative Ataxia Rating Scale (ICARS) and Scale for the Assessment and Rating of Ataxia (SARA) Scores With Face-to-Face and Tele-Assessment Methods in Ataxic Multiple Sclerosis Patients
Brief Title: Teleassessment in Ataxic Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, MSc physiotherapist, Hacettepe University
Other Study IDs: Tele-Assessment
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Ataxia; Multiple Sclerosis
MeSH Terms: conditions — Ataxia; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ataxic multiple sclerosis: In the study, those aged between 18-50 years, diagnosed with MS by a neurologist, Expanded Disability Status Scale (EDSS) score between 3-5, EDSS pyramidal system score ≤ 3 and cerebellar functional system score ≥ 1, patients who have been clinically stable for the last 3 months and have agreed to participate in the study will be included.

SUMMARY:
Our aim is to compare ICARS and SARA scores with face-to-face and tele-assessment methods in ataxic multiple sclerosis patients.

The hypotheses on which this study is based are; H1: Tele-assessment and face-to-face assessment results of the ICARS differ in patients with ataxic MS.

H2: Tele-assessment and face-to-face assessment results of SARA differ in patients with Ataxic MS.

DETAILED DESCRIPTION:
Patients will be evaluated both face-to-face and via tele-assessment (video conference call). In these evaluations, ICARS and SARA will be used. Face-to-face and tele-assessments will be applied on the same day, the order of administration will be decided by the randomization method, and a 10-minute rest will be given between the assessments.The interview will be recorded during the tele-assessment and a re-assessment will be made on the same recording 1 week later. Face-to-face assessment will be done as routinely done in the clinic. Face-to-face and tele-assessments will be made by 3 different assessors. Assessors will be blind to each other's assessment. All assessments will be carried out at Hacettepe University Faculty of Physical Therapy and Rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-50 years
* Being diagnosed with MS by a neurologist
* Expanded Disability Status Scale (EDSS) score between 3-5
* EDSS pyramidal system score ≤ 3 and cerebellar functional system score ≥ 1
* Being clinically stable for the last 3 months
* agree to participate in the study

Exclusion Criteria:

* Having other systemic, orthopedic or neurological disease
* Having a history of attacks in the last 3 months
* having peripheral vestibular complaints
* being mentally affected (Montreal Cognitive Rating Scale Score < 21)
* severe spasticity (Modified Ashworth Scale > 3)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ataxic MS patients with inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
ICARS | up to 6 months
  It will be used to assessment the severity of ataxia. ICARS consists of 4 sub-titles: posture and gait disorders, kinetic functions, speech disorders, and oculomotor disorders. The score range is in the range of 0-100, and higher scores indicate increased disease severity. It is a reliable and valid scale for ataxic MS patients. The assessment will take 20 minutes.
SARA | up to 6 months
  It will be used to assess the severity of ataxia. It is a scale that evaluates performance in 8 items as walking, standing, sitting, speech disorder, finger tracking, finger-nose test, rapid alternative hand movements, and heel-tibia test. The score range is 0-40, and an increase in the score indicates increased ataxia severity. It is a reliable and valid scale for ataxic MS patients. The assessment will take 15 minutes.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | up to 6 months
  Being between Expanded Disability Status Scale 3-5 and having a pyramidal system score below 3 are among the inclusion criteria. At the beginning of the study, all patients will be evaluated for EDSS, and patients who do not meet the criteria will not be included in the study. The assessment will take 15 minutes. The EDSS ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. EDSS steps 1.0 to 4.5 refer to people with MS who are able to walk without any aid. EDSS steps 5.0 to 9.5 are defined by the impairment to walking.
Montreal Cognitive Assessment (MoCA) | up to 6 months
  It will be used in the cognitive status assessment. Montreal Cognitive Assessment < 21 is among the exclusion criteria. At the beginning of the study, all patients will be given a MOCA, and patients who do not meet the criteria will not be included in the study. It assesses different cognitive dimensions including attention and concentration, executive functions, memory, language, visuospatial skills, abstract thinking, calculation, and orientation. The lowest score that can be obtained from the scale is 0, and the highest score is 30. Higher scores indicate a better cognitive levels. It is a reliable scale used for cognitive screening for MS patients. The assessment will take 10 minutes.
Telemedicine Satisfaction Questionnaire | up to 6 months
  It will be used to assess patients' satisfaction of the tele assessment method. After the tele-assesment is over, the questionnaire will be applied. The questionnaire consists of 14 items and patients are asked to rate each item from 1 to 5. The lowest score is 14 and the highest score is 70. A higher score indicates a higher level of satisfaction. It is a reliable and valid questionnaire for MS patients.
Telehealth Usability Questionnaire | up to 6 months
  It will be used to evaluate the usability of the teleassessment method by patients. After the tele-assesment is over, the questionnaire will be applied. The questionnaire consists of 21 items and patients are asked to rate each item from 1 to 7.The lowest score is 21 and the highest score is 147. A higher score indicates a higher level of usability. It is a reliable and valid questionnaire in MS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Kılınç, PhD, Study Director — Hacettepe University; Ender Ayvat, PhD, Principal Investigator — Hacettepe University; Fatma Ayvat, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)